CLINICAL TRIAL: NCT07406906
Title: The Effect of Dietary Supplements on Choroidal Thickness and Vasculature in Myopic Children: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Dietary Supplement for Myopia Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20251202005
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Myopia
Keywords: oral supplements, choroidal thickness, choroidal blood flow
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High concentration group (Experimental): 3 active capsules/ per day
  Interventions: Dietary Supplement: Oral dietary supplement provided in a capsule format (3 active capsules/ per day)
- Low-concentration group (Experimental): 1 active capsule and 2 placebo capsules/per day
  Interventions: Dietary Supplement: Oral dietary supplement provided in a capsule format (1 active capsule and 2 placebo capsules/per day)
- Control group (Placebo Comparator): 3 placebo capsules/per day
  Interventions: Other: Placebo control (3 placebo capsules/per day)

INTERVENTIONS:
Dietary Supplement: Oral dietary supplement provided in a capsule format (3 active capsules/ per day) — The active intervention in this study is an oral dietary supplement provided in a capsule format. The active ingredients include DHA/EPA and Astaxanthin.
  Arms: High concentration group
Dietary Supplement: Oral dietary supplement provided in a capsule format (1 active capsule and 2 placebo capsules/per day) — The active intervention in this study is an oral dietary supplement provided in a capsule format. The active ingredients include DHA/EPA and Astaxanthin.
  Arms: Low-concentration group
Other: Placebo control (3 placebo capsules/per day) — 3 placebo capsules/per day
  Arms: Control group

SUMMARY:
The purpose of this clinical trial is to investigate the changes in choroidal thickness and vasculature in myopic children following oral supplementation.

DETAILED DESCRIPTION:
Myopia commonly develops in childhood and is projected to affect nearly half of the global population by 2050, with high myopia posing a significant risk for irreversible vision loss. Although existing interventions can slow myopia progression, their use is limited by safety concerns, discomfort, variable efficacy, and accessibility, particularly in children. Therefore, exploring safe and accessible dietary oral supplements represents a promising alternative strategy for myopia control.

This study aims to conduct a 3-month, double-blind, placebo-controlled randomized clinical trial in myopic children to evaluate the effects of a specific dietary supplement on choroidal structure and vasculature and to explore its potential role in myopia control. The trial will compare changes in subfoveal and average choroidal thickness (ChT), choroidal vascularity index (CVI), axial length (AL), and spherical equivalent refraction (SER) among high-dose, low-dose, and placebo groups, assess the efficacy and safety of the combined supplementation. Subfoveal and average ChT, AL, visual acuity, cycloplegic SER, slit lamp, swept-source optical coherence tomography /angiography will be measured at 1-, 2-, and 3-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-13 years;
2. Cycloplegic spherical equivalent refraction (SER) of -0.50 D to -5.00 D with astigmatism of 2.5 D or less and best-corrected visual acuity (BCVA) of 0.0 logarithm or more in either eye;
3. Anisometropia of 1.50 D or less
4. Intraocular pressure of 10 mmHg to 21 mmHg in both eyes
5. Willing to give written consent to participate in the study and accept random allocation in grouping.

Exclusion Criteria:

1) Ocular abnormalities leading to visual impairment; 2) Severe physiological and psychological diseases affecting follow-up; 3) Receiving previous myopia control treatment including but not limited to atropine therapy and orthokeratology in the past 3 months; 4) Use of any other dietary supplements containing DHA/EPA, Lutein, or Astaxanthin in the past 3 months; 5) Known history of allergy to any of the components of the dietary supplement or placebo, or history of an allergic reaction that required emergency treatment; 6) Children who had other contraindications identified by the investigators that made them unsuitable for participation.

-

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in choroidal thickness measured by OCT | Choroidal thickness will be measured every month from enrollment to the end of treatment at 3 months.
  OCT and OCTA imaging will be performed using the swept-source OCT/OCTA system. ChT is defined as the perpendicular distance between the outer choroid-sclera margin and the retinal pigment epithelium-Bruch's complex. The average ChT and central ChT was calculated with the built-in software.

SECONDARY OUTCOMES:
Change in choroidal vasculature index | Choroidal vasculature index (CVI) will be measured every month from enrollment to the end of treatment at 3 months.
  OCT and OCTA imaging will be performed using the swept-source OCT/OCTA system. The average CVI and central CVI was calculated with the built-in software.
Change in axial length | Axial length will be measured every month from enrollment to the end of treatment at 3 months.
  Axial length, defined as the distance from the cornea to the retina, will be measured using an optical biometer. The average of three reliable measurements per eye will be recorded.
Change in cycloplegic spherical equivalent refraction | Spherical equivalent refraction will be measured every month from enrollment to the end of treatment at 3 months.
  Cycloplegia will be induced using a topical agent to temporarily paralyze the ciliary muscle. Refraction will then be measured using an autorefractor to determine the true Spherical Equivalent Refraction (SER).
Change in distance best-corrected visual acuity (BCVA) | BCVA will be measured every month from enrollment to the end of treatment at 3 months.
  BCVA will be measured using a visual chart at far distances.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No